CLINICAL TRIAL: NCT03179423
Title: Randomised, Double-Blind, Placebo-Controlled Study to Investigate GNbAC1 in Patients With Onset of Type 1 Diabetes Within 4 Years
Brief Title: Clinical Trial Assessing the GNbAC1 in Patients With Onset of Type 1 Diabetes Within 4 Years
Acronym: RAINBOW-T1D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GeNeuro Australia PTY Ltd (Industry)
Collaborators: Southern Star Research (Industry)
Responsible Party: Sponsor
Organization: GeNeuro SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNC-301
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Diabetes Mellitus, Type 1; T1D; Monoclonal antibody; Multiple Sclerosis associated retrovirus MSRV; Human Endogenous Retrovirus Type W (HERV-W); GNbAC1; Temelimab
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — temelimab

STUDY DESIGN:
Intervention Model Description: The first part of the trial is double-blind and the second part is open-label with all participants receiving the active treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNbAC1 (Experimental): Monthly IV repeated dose
  Interventions: Drug: GNbAC1
- Placebo (Placebo Comparator): Monthly IV repeated dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GNbAC1 — Monthly IV repeated dose
  Arms: GNbAC1
Drug: Placebo — Monthly IV repeated dose
  Arms: Placebo

SUMMARY:
The monoclonal antibody GNbAC1 targets the envelope protein (Env) of the human endogenous Multiple Sclerosis associated RetroVirus (MSRV), which could play a critical role in different autoimmune disorders, notably type 1 diabetes (T1D).

This study is a multicentre study evaluating for the first time the safety and efficacy of GNbAC1 in T1D subjects for a first bouble-blind period of 20 weeks followed by an optional open-label period of 24 weeks. The primary objective of the study is to assess the safety and tolerability of six consecutive 4-weekly doses of GNbAC1 in subjects with T1D. Secondary objectives are to determine the pharmacodynamic response to GNbAC1 on biomarkers of T1D.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects diagnosed with type 1 diabetes in the 4 years prior to signed informed consent;
* Peak stimulated C-peptide of ≥0.2 nmol/L during a mixed meal tolerance test performed during the Screening period;
* 18 to 55 years of age (both inclusive);
* Body weight >40 to ≤100 kg;
* Subjects positive for at least one diabetes-associated autoantibody (insulin, glutaminic-acid-decarboxylase-65 [GAD-65], tyrosine phosphatase-related antigen 2 [IA-2], ZnT8 or islet-cell antibody [ICA]).

Main Exclusion Criteria:

* Subjects with type 2 diabetes;
* Pregnant and nursing women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GNbAC1 in patients with recent onset type 1 diabetes: Serious Adverse Events (SAE) and Adverse Events (AE) | Week 1 to 24/48
  Serious Adverse Events (SAE) and Adverse Events (AE)

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (13):
  - Macquarie University Hospital, Macquarie University, New South Wales
  - AIM Centre, Merewether, New South Wales
  - Northern Sydney Local Health District - Royal North Shore Hospital, St Leonards, New South Wales
  - Ipswich Research Centre, Ipswich, Queensland
  - Mater Misericordiae Ltd and Mater Medical Research Institute Limited, South Brisbane, Queensland
  - Gold Coast Hospital and Health Service, Southport, Queensland
  - Southern Adelaide Local Health Network - Repatriation General Hospital, Adelaide, South Australia
  - Northern Adelaide Local Health Network Incorporated, operating as Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Eastern Health, Box Hill, Victoria
  - St Vincent's Hospital (Melbourne) Limited, Fitzroy, Victoria
  - Barwon Health - University of Geelong, Geelong, Victoria
  - Heidelberg Repatriation Hospital, Heidelberg, Victoria
  - Keogh Institute of Medical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No